CLINICAL TRIAL: NCT02957123
Title: Safety/Efficacy of Intranasally-Administered Bioactive Factors Produced by Autologous M2 Macrophages in Patients With Organic Brain Syndrome
Brief Title: Intranasal Inhalations of Bioactive Factors Produced by M2 Macrophages in Patients With Organic Brain Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alexander A Ostanin, Head of Clinical Department, Russian Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCI-25/05/2015
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Organic Brain Syndrome, Nonpsychotic; Neurocognitive Disorders; Mental Disorder, Organic; Delirium, Dementia, Amnestic, Cognitive Disorders; Nonpsychotic Organic Brain Syndrome; Organic Mental Disorder; Encephalopathy, Post-Traumatic, Chronic; Encephalopathy, Ischemic; Brain Ischemia
Keywords: macrophages M2 type; cytokines; intranasal administration; neuroprotection; neuroregeneration; organic brain syndrome; neurocognitive disorders
MeSH Terms: conditions — Neurocognitive Disorders; Chronic Traumatic Encephalopathy; Brain Ischemia

ARMS (1):
- Intranasal auto-M2-BFs (Experimental): Intranasally-Administered Bioactive Factors, Produced by Autologous M2 Macrophage (auto-M2-BFs). M2 macrophages were generated in vitro from peripheral blood of patients during 7 days.Cell-free culture medium, containing auto-M2-BFs, was collected and aliquots of 2 mL/vial were cryopreserved.
  30 patients with organic brain syndrome will receive auto-M2-BFs with the aerosol inhaler device (nebulizer), 2.0 mL once a day up to 30 days.
  Interventions: Drug: Intranasal auto-M2-BFs

INTERVENTIONS:
Drug: Intranasal auto-M2-BFs — Delivery is performed with the aerosol inhaler device (nebulizer), 2.0 mL once a day up to 30 days.
  Other Names: Bioactive Factors, Produced by M2 Macrophage

SUMMARY:
The investigators have designed an innovative proof-of-concept trial designed to provide data as to whether the treatment/rehabilitation efficacy and functional outcome of patients with organic brain syndrome are improved with intranasal inhalations of bioactive factors (BF), produced by autologous M2 macrophages (auto-M2-BFs). The rationale for this approach is the ability of central nervous system to repair and the important role of macrophages in the regulation of this process. It was found that type 2 macrophages have anti-inflammatory and reparative potential, whereas M1 cells possess pro-inflammatory and neurotoxic effects. Action of M2 macrophages is largely realized through the production a wide variety of bioactive factors (cytokines, chemokines, growth factors, neuropeptides, microvesicles etc) that inhibit inflammation, protect neurons from apoptosis, stimulate neurogenesis, the growth and remyelination of axons, the formation of new synapses and activate angiogenesis. This study uses auto-M2-BFs, as therapeutic agents and intranasal administration focusing on nose to brain transport, as a mode of delivery. Expected clinical effects in treated subjects: improvement of cognitive functions (memory, language, attention); correction of focal neurological deficit (paresis, spasticity, sensory disorders); reduction vestibular/ataxic disorders (vertigo, unsteadiness when walking); reduction of headaches; reduction of asthenia (weakness, fatigue); correction of emotional disorders (anxiety, depression).

DETAILED DESCRIPTION:
Following injury to the central nervous system (CNS), immune-mediated inflammation profoundly affects the ability of neural cells to survive and to regenerate. The role of inflammation comprises mostly of macrophages, is controversial, since macrophages can both induce neuronal and glial toxicity and promote tissue repair. The opposite effects of macrophages may be conditioned by their functional heterogeneity. Thus, classical pro-inflammatory macrophages (M1) are tissue-destructive, while anti-inflammatory (M2) macrophages mediate tissue repair. In addition, M2 macrophages predominantly induce the Th2 response, which is particularly beneficial in CNS repair. Using low serum conditions the investigators have generated M2-like macrophages and evaluated their phenotypic and functional features [1, 2]. Our data indicate that M2 macrophages, in contrast to pro-inflammatory M1 cells, produced significantly lower levels of pro-inflammatory cytokines (IL-1β, tumor necrosis factor-α, IL-6, IL-18, IL-12), chemokines (IL-8, monocyte chemoattractant protein 1-1) and Th1/Th2-cytokines (interferon-γ, IL-2, IL-4) coupled with a higher IL-10 level. M2 macrophages were capable of producing neurotrophic- (brain-derived neurotrophic factor,insulin-like growth factor-1), angiogenic- (vascular endothelial growth factor), and other growth factors (erythropoietin, granulocyte-colony stimulating factor , basic fibroblast growth factor, epidermal growth factor) with neuroprotective and regenerative activity.

Our pilot clinical trials have demonstrated the safety and clinical efficacy of intrathecal administration of M2 macrophages in children with severe cerebral palsy [3] and in non-acute stroke patients [4].

Since cell-free culture medium of M2 macrophages contains a wide variety of neurotrophic, immunoregulatory and pro-angiogenic factors, the investigators expect that intranasal administration of these auto-M2-BFs will improve the treatment/rehabilitation efficacy and functional outcome of patients with organic brain syndrome. Of note, intranasal administration of M2-macrophage soluble factors allow to delivery bioactive agents to brain through the olfactory and trigeminal ways across brain-blood barrier.

ELIGIBILITY:
Inclusion Criteria:

* Adults: age 18 - 80
* Persistent neurological deficits (cognitive, mental, motor, vestibular/ataxic disorders as a result of trauma, cardiovascular, neurodegenerative and others cerebral injuries), confirmed clinically and by CT or MRI
* A written informed consent of the patient or close relatives

Exclusion Criteria:

* Psychiatric disorders
* Seizures
* Severe dementia
* Hepatic or renal dysfunctions
* Hemodynamic or respiratory instability
* HIV or uncontrolled bacterial, fungal, or viral infections
* Pregnancy
* Malignancy
* Intolerance to gentamicin and / or multiple drug allergies
* Participation in other clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena R Chernykh, MD, PhD, Study Chair — Institute of Fundamental and Clinical Immunology; Alexander A Ostanin, MD, PhD, Principal Investigator — Institute of Fundamental and Clinical Immunology
Locations (1):
- Institute of Fundamental and Clinical Immunology, Novosibirsk, Russia

REFERENCES:
- [Background] Chernykh ER, Shevela EY, Sakhno LV, Tikhonova MA, Petrovsky YL, Ostanin AA. The generation and properties of human M2-like macrophages: potential candidates for CNS repair? Cell Ther Transplant., 2010 DOI: 10.3205/ctt-2010-en-000080.01
- [Background] Sakhno LV, Shevela EY, Tikhonova MA, Ostanin AA, Chernykh ER. The Phenotypic and Functional Features of Human M2 Macrophages Generated Under Low Serum Conditions. Scand J Immunol. 2016 Feb;83(2):151-9. doi: 10.1111/sji.12401. PMID 26678544
- [Background] Chernykh ER, Kafanova MY, Shevela EY, Sirota SI, Adonina EI, Sakhno LV, Ostanin AA, Kozlov VV. Clinical experience with autologous M2 macrophages in children with severe cerebral palsy. Cell Transplant. 2014;23 Suppl 1:S97-104. doi: 10.3727/096368914X684925. Epub 2014 Oct 9. PMID 25302537
- [Background] Chernykh ER, Shevela EY, Starostina NM, Morozov SA, Davydova MN, Menyaeva EV, Ostanin AA. Safety and Therapeutic Potential of M2 Macrophages in Stroke Treatment. Cell Transplant. 2016;25(8):1461-71. doi: 10.3727/096368915X690279. Epub 2015 Dec 14. PMID 26671426
- [Result] Shevela EY., Davydova MN, Starostina NM, Yankovskaya AA, Ostanin AA, Chernykh ER. Intranasal delivery of M2 macrophage-derived soluble products reduces neurological deficit in patients with cerebrovascular disease: A Pilot Study. Journal of Neurorestoratology, 2019; 7: 89-100 doi:10.26599/JNR.2019.9040010

RESULTS

PARTICIPANT FLOW:
Groups:
- Intranasal Auto-M2-BFs: Intranasally-Administered Bioactive Factors (BF), Produced by Autologous M2 Macrophage (auto-M2-BFs). 30 patients with organic brain syndrome will receive auto-M2-BFs as intranasal inhalations with the aerosol inhaler device (nebulizer), 2.0 mL once a day up to 30 days.
Period: Overall Study
Arm/Group | Intranasal Auto-M2-BFs
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 30 patients (male and female; 18-80 years old; from Russia) with organic brain syndrome
Groups:
- Intranasal Auto-M2-BFs: Intranasally-Administered Bioactive Factors, Produced by Autologous M2 Macrophage (auto-M2-BFs). 30 patients with organic brain syndrome will receive auto-M2-BFs as intranasal inhalations with the aerosol inhaler device (nebulizer), 2.0 mL once a day up to 30 days.
Arm/Group | Intranasal Auto-M2-BFs
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 30

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Severe Adverse Events and Adverse Reactions
Description: Occurrence of severe adverse events and adverse reactions (allergic, toxic, inflammatory reactions; neurological deterioration, convulsive syndrome)
Time Frame: up to 6 months after treatment
Population: The number of patients with severe adverse events and adverse reactions
Measure: Count of Participants; unit: Participants
Groups:
- Intranasal Auto-M2-BFs: Intranasally-Administered Bioactive Factors, Produced by Autologous M2 Macrophage (auto-M2-BFs). M2 macrophages were generated in vitro from peripheral blood of patients during 7 days.Cell-free culture medium, containing auto-M2-BFs, was collected and aliquots of 2 mL/vial were cryopreserved.
  30 patients with organic brain syndrome will receive their first doses (n=2-3) of auto-M2-BFs in clinic and wait 2 hrs to determine any short-time adverse effects of inhaled dose.
  The subsequent course of intranasal inhalations (once a day up to 30 days) performed as outpatient treatment.
  Intranasal auto-M2-BFs: Delivery is performed with the aerosol inhaler device (nebulizer), 2.0 mL once a day up to 30 days.
Arm/Group | Intranasal Auto-M2-BFs
Number analyzed (Participants) | 30
Participants | 0

2. Secondary Outcome: Change in Subjective Assessment of Clinical Symptoms (SACS)
Description: Subjective Assessment of Clinical Symptoms (SACS) is a 5-point rating scale with standardized criteria (0 - no; 1 - mild; 2 - moderate; 3 - severe; 4 - intensive) subjective assessment of the severity of fifteen clinical symptoms most characteristic of neurological disorders (headache, dizziness, gait disturbance, speech, visual impairment, tremor et al). Minimum SACS "total" score is 0, and maximum SACS "total" score is 60. Neurological improvements are assessed by SACS "total" score as > 6 points' reduction from baseline.
Time Frame: Baseline and 6 months after treatment
Population: Patients with neurological improvements are assessed by SACS "total" score as > 6 points' reduction from baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Intranasal Auto-M2-BFs
Number analyzed (Participants) | 30
Participants | 12

3. Secondary Outcome: Change in Hospital Anxiety and Depression Scale (HADS)
Description: Hospital Anxiety and Depression Scale (HADS) is used to diagnose anxiety/depression symptoms (absence - 0~7 points; subclinical form - 8~10 points; clinical form - 11 points or more). Minimum HADS "total" score (anxiety + depression subscale) is 0, and maximum HADS "total" score is 42. Improvements in patients with anxiety/depression symptoms are assessed by HADS "total" score as > 4 points reduction from baseline.
Time Frame: Baseline and 6 months after treatment
Population: Improvements in patients with anxiety/depression symptoms are assessed by HADS "total" score as > 4 points reduction from baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Intranasal Auto-M2-BFs
Number analyzed (Participants) | 26
Participants | 14

4. Secondary Outcome: Change in Functional Mobility Assessment (FMA) Scale
Description: Functional Mobility Assessment (FMA) iscale is designed to evaluate parameters characterizing stability (0~24 points) and gait (0~16 points).
  The maximum FMA "total" score on stability and gait subscales is 39-40 and corresponds to the norm, minimum FMA "total" score is 0 and corresponds to the gross impairment. The degree of impairment of "total" score is divided into significant (0~20 points), moderate (21~33 points), and light (34~38 points), whereas 39~40 points indicate no impairments. Improved mobility is assessed as FMA "total" score enhancement > 4 points from baseline.
Time Frame: Baseline and 6 months after treatment
Population: Improved mobility is assessed as FMA "total" score enhancement > 4 points from baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Intranasal Auto-M2-BFs
Number analyzed (Participants) | 28
Participants | 16

5. Secondary Outcome: Change in Montreal Cognitive Assessment (МоСА)
Description: Montreal Cognitive Assessment (MoCa) is used to assess cognitive functions. The maximum MoCa "total" score is 26-30 points and corresponds to the norm, 19-25 points - mild cognitive disorder; 11-21 points - dementia. Improvements in patients with cognitive disorder are assessed as MoCA "total" score increase > 3 points from baseline.
Time Frame: Baseline and 6 months after treatment
Population: Improvements in patients with cognitive disorder are assessed as MoCA MoCA "total" score increase > 3 points from baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Intranasal Auto-M2-BFs
Number analyzed (Participants) | 19
Participants | 10

ADVERSE EVENTS:
Time Frame: The severe adverse events and adverse reactions (allergic, toxic, inflammatory reactions; neurological deterioration, convulsive syndrome) were collected up to 6 months after treatment
Arm/Group | Intranasal Auto-M2-BFs
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2015-10-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT02957123/Prot_000.pdf
  • Informed Consent Form (2015-10-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT02957123/ICF_001.pdf
  • Statistical Analysis Plan (2015-10-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT02957123/SAP_002.pdf